CLINICAL TRIAL: NCT04865159
Title: A Phase I, Open-label Clinical Pharmacology Study to Evaluate the Effect of Tipifarnib on Cardiac Safety in Subjects With Advanced Solid Malignancies
Brief Title: Cardiovascular Safety Study of Tipifarnib in Patients With Advanced Solid Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated due to recruitment challenges
Sponsor: Kura Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: KO-TIP-011
Expanded Access: NCT04809233 (Available)
Record Dates: First submitted 2021-03-04; First posted 2021-04-29 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-04

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — tipifarnib

STUDY DESIGN:
Intervention Model Description: Tipifarnib will be administered with a meal at a starting single dose of 900 mg, orally, once on Day 1, Cycle 1 followed by 600 mg, orally bid on Cycle 1 Days 2-7 and Days 15-21 for a 28-day treatment cycle.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Group Assignment (Other): Single Arm - Drug administered on Days 1-7 and Days 15-21 of a 28-day treatment cycle. Series of Pharmacokinetics and ECGs will be done during cycle 1.
  Interventions: Drug: Tipifarnib

INTERVENTIONS:
Drug: Tipifarnib — Cardiac Safety of Tipifarnib

SUMMARY:
A Phase I, open-label clinical pharmacology study designed to evaluate the effect of tipifarnib on cardiac repolarization (corrected QT interval [QTc] duration) following a single dose of 900 mg and after repeated twice daily administration of 600 mg in subjects with advanced solid malignancies. Subjects will receive a 900 mg single dose at cycle 1 day 1 follow by 600 mg twice a day orally with a meal (Days 2-7 and 15-21) in 28-day cycles. Beginning on Day 2 of Cycle 1, subjects will self-administer 600 mg tipifarnib, orally with a meal, bid for 7 days in alternating weeks (Days 2-7 and 15-21) in 28-day cycles. The secondary objectives are to evaluate the safety and PK of tipifarnib. Series of PK will be collected on day -1 of Cycle 1, Cycle 1 day 1 and Cycle 1 day 7.

DETAILED DESCRIPTION:
Phase I study will evaluate the effect of tipifarnib on cardiac repolarization (corrected QT interval [QTc] duration) following a single dose of 900 mg and after repeated twice daily administration of 600 mg in subjects with advanced solid malignancies. The study will enroll approximately 20 subjects with advanced solid malignancies (at least 8, but no more than 12, male subjects). Subjects must have no approved/appropriate therapeutic options available. Subject will undergo series of ECG at Cycle 1 day -1 follow by study drug dosing, series of Pharmacokinetic and ECG at Cycle 1 day 1 and Cycle 1 day 7. Beginning on Day 2 of Cycle 1, subjects will self-administer 600 mg tipifarnib, orally with a meal, bid for 7 days in alternating weeks (Days 2-7 and 15-21) in 28-day cycles. For Cycle 2 and beyond, subjects will self-administer 600 mg bid on Days 1-7 and Days 15-21 in 28-day cycles.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age.
2. Advanced solid tumor malignancies for whom no other therapy or intervention is available
3. Confirmation of measurable disease by RECIST v1.1
4. No uncontrolled hypertension, defined as >140/90 mm Hg
5. A normal 12-lead ECG
6. At least two weeks since the last systemic anticancer therapy regimen prior to Cycle 1 Day 1; this includes radiation therapy.
7. ECOG performance status of 0-2.
8. Acceptable liver, renal and hematological function
9. Other protocol defined inclusion criteria may apply.

Exclusion Criteria

1. Has disease that is suitable for therapy administered with curative intent.
2. Ongoing treatment with another anticancer agent indicated for the malignancy for which the subject is enrolling into the study (excluding adjuvant hormonal therapy for breast cancer and hormonal treatment for castration sensitive prostate cancer).
3. History of cardiomyopathy, unstable angina within prior 6 months, myocardial infarction within prior 6 months, cerebrovascular attack within prior 6 months, history of New York Heart Association grade III or greater congestive heart failure, or current serious cardiac arrhythmia requiring medication.
4. Non-tolerable Grade 2 or ≥ Grade 3 neuropathy or evidence of unstable neurological symptoms within 4 weeks of Cycle 1 Day 1.
5. Major surgery, other than diagnostic surgery, within 14 days prior to Cycle 1 Day 1, without complete recovery.
6. Active, uncontrolled bacterial, viral or fungal infections requiring systemic therapy.
7. Other protocol defined exclusion may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-05-02 (Actual)

PRIMARY OUTCOMES:
The change from baseline in time-matched difference in QTc interval to post-baseline time points after a single 900 mg dose and multiple 600 mg BID doses of tipifarnib in subjects with Advanced Solid Malignancies | 7 days
  The analysis will be performed using the concentration-QTc modeling approach (Garnett 2018) and the by-time point modeling approach defined in the International Council on Harmonisation (ICH) E14 guidance. The analysis will be performed using triplicate, time-matched ECG measurements of the QTc interval will be taken at baseline, Day 1 (900 mg tipifarnib) and Day 7 (600 mg tipifarnib BID) at predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours post dose (24 hour on day 1 only).

SECONDARY OUTCOMES:
Investigate safety and tolerability of tipifarnib according to NCI CTCAE v5.0 | 30 days after treatment discontinuation
  Incidence of adverse events, incidence of abnormal laboratory test results, abnormal vital signs, and abnormal ECG results

CONTACTS AND LOCATIONS:
Overall Officials: David Sommerhalder, MD, Principal Investigator — NEXT Oncology
Locations (3):
- United States (3):
  - Gabrail Cancer Center Research, Canton, Ohio
  - NEXT Oncology, Austin, Texas
  - NEXT Oncology, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No